CLINICAL TRIAL: NCT00002925
Title: Phase I Study of MDR Modulation With PSC-833 (NSC# 648265) With a Pilot Study of Cytogenetic Risk-Adapted Consolidation Followed by a Phase II Pilot Study of Immunotherapy With RIL-2 (NSC # 373364) in Previously Untreated Patients With AML< 60 Years
Brief Title: Combination Chemotherapy Plus PSC 833 Followed by Interleukin-2 in Treating Patients With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Monica M Bertagnolli, MD, Cancer and Leukemia Group B
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065333; U10CA031946 (NIH); CLB-9621
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2011-03

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Cytarabine; Daunorubicin; Etoposide; valspodar; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADE (Active Comparator)
  Interventions: Drug: ara-C; Drug: Daunorubicin; Drug: Etoposide; Biological: Aldesleukin
- ADEP (Experimental)
  Interventions: Drug: ara-C; Drug: Daunorubicin; Drug: Etoposide; Drug: PSC-833; Biological: Aldesleukin

INTERVENTIONS:
Drug: ara-C
Drug: Daunorubicin
Drug: Etoposide
Drug: PSC-833
  Arms: ADEP
Biological: Aldesleukin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Some cancers may become resistant to chemotherapy drugs. Combining PSC 833 with chemotherapy may reduce resistance to the drugs and allow the cancer cells to be killed. Interleukin-2 may stimulate a person's white blood cells to kill leukemia cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy plus PSC 833 followed by additional chemotherapy or peripheral stem cell transplantation and interleukin-2 in treating patients with untreated acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of daunorubicin when used in combination with etoposide, cytarabine, and PSC 833 (ADEP), and in combination with etoposide and cytarabine (ADE) in previously untreated patients with acute myelogenous leukemia who are less than 60 years. II. Determine the MTD of etoposide when used in combination with a constant dose of daunorubicin and cytarabine (ADE) in these patients. III. Determine the feasibility and toxic effects of administering postremission therapy in a risk adapted fashion, such that patients with favorable cytogenetic findings receive three intensifications with high dose cytarabine (HiDAC), while average to poor risk patients receive HiDAC/etoposide/filgrastim (G-CSF) for consolidation therapy and stem cell mobilization followed by peripheral stem cell (PBSC) transplant using busulfan/etoposide as the preparative regimen. IV. Determine the feasibility and toxic effects of the consolidation sequence of HiDAC/etoposide/G-CSF followed by 2 courses of HiDAC in patients who would otherwise receive PBSC transplant, but are unable to do so for logistical or institutional reasons. V. Determine the feasibility of intermittent administration of high dose subcutaneous interleukin-2 (IL-2) in combination with continuous low dose subcutaneous IL-2 in patients recovering from PBSC transplant or intensive consolidation chemotherapy.

OUTLINE: This is a dose escalation study of daunorubicin in the induction therapy portion, with a separate dose escalation study of etoposide in the same portion. Patients are treated with three phases of treatment: induction, intensification, and postremission therapy. Induction therapy: Patients receive cytarabine IV as a continuous infusion on days 1-7 plus daunorubicin IV over 30 minutes and etoposide IV over 2 hours on days 1-3 (ADE regimen). Some patients also receive PSC 833 IV as a continuous infusion on days 1-3 (ADEP regimen). This course may be repeated 14 days later. Cohorts of 9 patients each receive escalating doses of daunorubicin until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose at which 3 of 9 patients experience dose limiting toxicity. Escalations are conducted separately for the ADE and ADEP regimens. Other cohorts of 9 patients each receive escalating doses of etoposide with constant doses of daunorubicin in the ADE regimen. The MTD is described in the same manner. Intensification therapy: Arm I (patients with certain genetic characteristics in their leukemia cells): Patients receive 3 additional courses of cytarabine IV over 3 hours, twice a day, for 3 days. Courses are repeated every 28 days. Arm II (patients who do not have these genetic characteristics): Patients undergo a peripheral blood stem cell (PBSC) transplant. Patients first receive high dose cytarabine IV over 2 hours on days 1-4, etoposide IV as a continuous infusion on days 1-4, and filgrastim (G-CSF) subcutaneously beginning on day 5 until blood counts recover. PBSC are then collected. Approximately 4-6 weeks later, patients receive oral busulfan 4 times a day on days 1-4 and etoposide IV over 4 hours on day 5. PBSC are reinfused on day 7. G-CSF is administered subcutaneously beginning on day 7 until blood cell counts recover. Arm III (patients who cannot undergo a PBSC transplant): Patients receive cytarabine, etoposide, and G-CSF as in arm II, then high dose cytarabine as in arm I. Postremission therapy (all patients): Patients receive low dose interleukin-2 (IL-2) by daily injection for 2 weeks. On day 15, patients begin receiving intermittent high dose IL-2 three days a week. Patients alternate these courses of IL-2: 14 days of low dose IL-2, 3 days of high dose IL-2, 1 day of rest, low dose IL-2 for 10 days, then 3 days of high dose IL-2, then 1 day of rest. This course is repeated 3 times. Patients then receive another 16 day course of low dose IL-2. Patients are followed at 1 month, then every 3 months for 2 years, then every 6 months for 2 years, then annually thereafter.

PROJECTED ACCRUAL: Approximately 410 patients will be accrued into this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven acute myelogenous leukemia, except M3

PATIENT CHARACTERISTICS: Age: 15 to 59 Performance status: Not specified Life expectancy: Not specified Hematopoietic: No prior hematologic malignancy, myeloproliferative disorder, myelodysplastic syndrome, or paroxysmalnocturnal hemoglobinuria No unexplained cytopenias greater than 3 months in duration Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy No prior treatment for leukemia except leukapheresis Chemotherapy: No prior chemotherapy except hydroxyurea which may be used for emergency therapy of hyperleukocytosis Endocrine therapy: Not specified Radiotherapy: Prior cranial radiation therapy allowed for CNS leukostasis Surgery: Not specified

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 410 (Actual)
Dates: Start 1997-02; Primary Completion 2003-11 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E. Kolitz, MD, Study Chair — Don Monti Comprehensive Cancer Center at North Shore University Hospital
Locations (33):
- United States (33):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Background] Langer C, Maharry K, Mrózek K, et al.: Low Meningioma 1 (MN1) gene expression to predict outcome in cytogenetically normal acute myeloid leukemia (CN-AML): A Cancer and Leukemia Group B (CALGB) study. [Abstract] J Clin Oncol 26 (Suppl 15): A-7011, 2008.
- [Background] Langer C, Radmacher MD, Ruppert AS, Whitman SP, Paschka P, Mrozek K, Baldus CD, Vukosavljevic T, Liu CG, Ross ME, Powell BL, de la Chapelle A, Kolitz JE, Larson RA, Marcucci G, Bloomfield CD; Cancer and Leukemia Group B (CALGB). High BAALC expression associates with other molecular prognostic markers, poor outcome, and a distinct gene-expression signature in cytogenetically normal patients younger than 60 years with acute myeloid leukemia: a Cancer and Leukemia Group B (CALGB) study. Blood. 2008 Jun 1;111(11):5371-9. doi: 10.1182/blood-2007-11-124958. Epub 2008 Mar 31. PMID 18378853
- [Background] Marcucci G, Maharry K, Radmacher MD, Mrozek K, Vukosavljevic T, Paschka P, Whitman SP, Langer C, Baldus CD, Liu CG, Ruppert AS, Powell BL, Carroll AJ, Caligiuri MA, Kolitz JE, Larson RA, Bloomfield CD. Prognostic significance of, and gene and microRNA expression signatures associated with, CEBPA mutations in cytogenetically normal acute myeloid leukemia with high-risk molecular features: a Cancer and Leukemia Group B Study. J Clin Oncol. 2008 Nov 1;26(31):5078-87. doi: 10.1200/JCO.2008.17.5554. Epub 2008 Sep 22. PMID 18809607
- [Background] Paschka P, Marcucci G, Ruppert AS, Whitman SP, Mrozek K, Maharry K, Langer C, Baldus CD, Zhao W, Powell BL, Baer MR, Carroll AJ, Caligiuri MA, Kolitz JE, Larson RA, Bloomfield CD. Wilms' tumor 1 gene mutations independently predict poor outcome in adults with cytogenetically normal acute myeloid leukemia: a cancer and leukemia group B study. J Clin Oncol. 2008 Oct 1;26(28):4595-602. doi: 10.1200/JCO.2007.15.2058. Epub 2008 Jun 16. PMID 18559874
- [Background] Marcucci G, Maharry K, Whitman SP, Vukosavljevic T, Paschka P, Langer C, Mrozek K, Baldus CD, Carroll AJ, Powell BL, Kolitz JE, Larson RA, Bloomfield CD; Cancer and Leukemia Group B Study. High expression levels of the ETS-related gene, ERG, predict adverse outcome and improve molecular risk-based classification of cytogenetically normal acute myeloid leukemia: a Cancer and Leukemia Group B Study. J Clin Oncol. 2007 Aug 1;25(22):3337-43. doi: 10.1200/JCO.2007.10.8720. Epub 2007 Jun 18. PMID 17577018
- [Background] Metzeler KH, Hummel M, Bloomfield CD, et al.: An 86-probe gene expression signature can predict survival in AML with normal karyotype independently of FLT3 ITD and NPM1 mutation status: a collaborative study from the AMLCG and CALGB study groups. [Abstract] Blood 110 (11): A-596, 2007.
- [Background] Whitman SP, Ruppert AS, Marcucci G, Mrozek K, Paschka P, Langer C, Baldus CD, Wen J, Vukosavljevic T, Powell BL, Carroll AJ, Kolitz JE, Larson RA, Caligiuri MA, Bloomfield CD. Long-term disease-free survivors with cytogenetically normal acute myeloid leukemia and MLL partial tandem duplication: a Cancer and Leukemia Group B study. Blood. 2007 Jun 15;109(12):5164-7. doi: 10.1182/blood-2007-01-069831. Epub 2007 Mar 6. PMID 17341662
- [Background] Paschka P, Marcucci G, Ruppert AS, Mrozek K, Chen H, Kittles RA, Vukosavljevic T, Perrotti D, Vardiman JW, Carroll AJ, Kolitz JE, Larson RA, Bloomfield CD; Cancer and Leukemia Group B. Adverse prognostic significance of KIT mutations in adult acute myeloid leukemia with inv(16) and t(8;21): a Cancer and Leukemia Group B Study. J Clin Oncol. 2006 Aug 20;24(24):3904-11. doi: 10.1200/JCO.2006.06.9500. PMID 16921041
- [Background] Kolitz JE, George SL, Baer MR, Lee EJ, Bloomfield CD, Larson RA; Cancer and Leukemia Group B (CALGB) trials in younger and older adults. P-glycoprotein (Pgp) modulation in untreated acute myeloid leukemia (AML): Cancer and Leukemia Group B (CALGB) trials in younger and older adults. Ann Hematol. 2004;83 Suppl 1:S103-4. doi: 10.1007/s00277-004-0850-2. No abstract available. PMID 15124695
- [Background] Sekeres MA, Peterson B, Dodge RK, Mayer RJ, Moore JO, Lee EJ, Kolitz J, Baer MR, Schiffer CA, Carroll AJ, Vardiman JW, Davey FR, Bloomfield CD, Larson RA, Stone RM; Cancer and Leukemia Group B. Differences in prognostic factors and outcomes in African Americans and whites with acute myeloid leukemia. Blood. 2004 Jun 1;103(11):4036-42. doi: 10.1182/blood-2003-09-3118. Epub 2004 Feb 19. PMID 14976037
- [Background] Sekeres MA, Dodge RK, Bloomfield CD, et al.: Racial differences in prognostic factors and outcome in acute myeloid leukemia (AML): a Cancer and Leukemia Group B (CALGB) study. [Abstract] Blood 100 (11 Pt 1): A-323, 2002.
- [Result] Radmacher MD, Marcucci G, Ruppert AS, Mrozek K, Whitman SP, Vardiman JW, Paschka P, Vukosavljevic T, Baldus CD, Kolitz JE, Caligiuri MA, Larson RA, Bloomfield CD; Cancer and Leukemia Group B. Independent confirmation of a prognostic gene-expression signature in adult acute myeloid leukemia with a normal karyotype: a Cancer and Leukemia Group B study. Blood. 2006 Sep 1;108(5):1677-83. doi: 10.1182/blood-2006-02-005538. Epub 2006 May 2. PMID 16670265
- [Result] Marcucci G, Baldus CD, Ruppert AS, et al.: Overexpression of the ERG gene is an adverse prognostic factor in acute myeloid leukemia (AML) with normal cytogenetics (NC): a Cancer and Leukemia Group B study (CALGB). [Abstract] Blood 106 (11): A-335, 2005.
- [Result] Marcucci G, Baldus CD, Ruppert AS, Radmacher MD, Mrozek K, Whitman SP, Kolitz JE, Edwards CG, Vardiman JW, Powell BL, Baer MR, Moore JO, Perrotti D, Caligiuri MA, Carroll AJ, Larson RA, de la Chapelle A, Bloomfield CD. Overexpression of the ETS-related gene, ERG, predicts a worse outcome in acute myeloid leukemia with normal karyotype: a Cancer and Leukemia Group B study. J Clin Oncol. 2005 Dec 20;23(36):9234-42. doi: 10.1200/JCO.2005.03.6137. Epub 2005 Nov 7. PMID 16275934
- [Result] Marcucci G, Radmacher MD, Ruppert AS, et al.: Independent validation of prognostic relevance of a previously reported gene-expression signature in acute myeloid leukemia (AML) with normal cytogenetics (NC): a Cancer and Leukemia Group B (CALGB) study. [Abstract] Blood 106 (11): A-755, 2005.
- [Result] Kolitz JE, George SL, Dodge RK, Hurd DD, Powell BL, Allen SL, Velez-Garcia E, Moore JO, Shea TC, Hoke E, Caligiuri MA, Vardiman JW, Bloomfield CD, Larson RA; Cancer and Leukemia Group B. Dose escalation studies of cytarabine, daunorubicin, and etoposide with and without multidrug resistance modulation with PSC-833 in untreated adults with acute myeloid leukemia younger than 60 years: final induction results of Cancer and Leukemia Group B Study 9621. J Clin Oncol. 2004 Nov 1;22(21):4290-301. doi: 10.1200/JCO.2004.11.106. PMID 15514371
- [Result] Baldus CD, Tanner SM, Ruppert AS, Whitman SP, Archer KJ, Marcucci G, Caligiuri MA, Carroll AJ, Vardiman JW, Powell BL, Allen SL, Moore JO, Larson RA, Kolitz JE, de la Chapelle A, Bloomfield CD. BAALC expression predicts clinical outcome of de novo acute myeloid leukemia patients with normal cytogenetics: a Cancer and Leukemia Group B Study. Blood. 2003 Sep 1;102(5):1613-8. doi: 10.1182/blood-2003-02-0359. Epub 2003 May 15. PMID 12750167
- [Result] Kolitz JE, George SL, Barrier R, et al.: Treatment of core binding factor (CBF) acute myeloid leukemia (AML) with post-remission high-dose cytarabine (HiDAC): results from CALGB 9621. [Abstract] Blood 102 (11 Pt 1): A-612, 2003.
- [Result] Kolitz JE, George SL, Barrier R, et al.: A novel post-remission consolidation regimen for patients with acute myeloid leukemia (AML) < 60 years old with normal or unfavorable cytogenetics: results from CALGB 9621. [Abstract] Blood 102 (11 Pt 1): A-609, 2003.
- [Result] Mrozek K, Prior TW, Edwards C, Marcucci G, Carroll AJ, Snyder PJ, Koduru PR, Theil KS, Pettenati MJ, Archer KJ, Caligiuri MA, Vardiman JW, Kolitz JE, Larson RA, Bloomfield CD. Comparison of cytogenetic and molecular genetic detection of t(8;21) and inv(16) in a prospective series of adults with de novo acute myeloid leukemia: a Cancer and Leukemia Group B Study. J Clin Oncol. 2001 May 1;19(9):2482-92. doi: 10.1200/JCO.2001.19.9.2482. PMID 11331327
- [Result] Whitman SP, Archer KJ, Feng L, Baldus C, Becknell B, Carlson BD, Carroll AJ, Mrozek K, Vardiman JW, George SL, Kolitz JE, Larson RA, Bloomfield CD, Caligiuri MA. Absence of the wild-type allele predicts poor prognosis in adult de novo acute myeloid leukemia with normal cytogenetics and the internal tandem duplication of FLT3: a cancer and leukemia group B study. Cancer Res. 2001 Oct 1;61(19):7233-9. PMID 11585760
- [Result] Kolitz JE, George SL, Hurd D, et al.: Parallel phase I trials of multi-drug resistance (MDR) modulation with PSC-833 in untreated patients (PTS) with acute myeloid leukemia (AML) less than 60 years old: preliminary results of CALGB 9621. Blood 94(suppl 1): A-1705, 384a, 1999.
- [Result] Kolitz JE, Georg SL, Hurd D, et al.: Cytogenetic risk-adapted intensification followed by immunotherapy with recombinant interleukin-2 (rIL-2) in patients (PTS) less than 60 years old with acute myeloid leukemia (AML) in first complete remission (CR): preliminary results of CALGB 9621. Blood 94(suppl 1): A-2582, 579a, 1999.